CLINICAL TRIAL: NCT02082470
Title: Feasibility and Preliminary Outcomes of Survivorship Care Planning in Ovarian Cancer
Brief Title: Survivorship Care Planning in Improving Quality of Life in Survivors of Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14001; NCI-2014-00423 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 14001 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2014-03-06; First posted 2014-03-10 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-09

CONDITIONS: Cancer Survivor; Stage IA Ovarian Epithelial Cancer; Stage IB Ovarian Epithelial Cancer; Stage IC Ovarian Epithelial Cancer; Stage IIA Ovarian Epithelial Cancer; Stage IIB Ovarian Epithelial Cancer; Stage IIC Ovarian Epithelial Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIC Ovarian Epithelial Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Aftercare; Watchful Waiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (standard post-treatment) (Active Comparator): Participants receive standard post-treatment care consisting of regular cancer surveillance visits with treating oncologists.
  Interventions: Other: active surveillance; Other: questionnaire administration
- Arm II (survivorship care planning) (Experimental): Participants complete survivorship care planning in close collaboration with treating oncologists.
  Interventions: Other: follow-up care; Other: questionnaire administration

INTERVENTIONS:
Other: follow-up care — Undergo survivorship care planning
  Arms: Arm II (survivorship care planning)
Other: active surveillance — Undergo cancer surveillance
  Arms: Arm I (standard post-treatment)
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies survivorship care planning in supporting quality of life in ovarian cancer survivors following primary treatment. Survivorship care plans have the potential to empower patients and provide them with a plan of care following treatments. Survivorship care planning may support patient's overall well-being and quality of life after treatment of ovarian cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and acceptability of survivorship care planning (SCP) in ovarian cancer.

SECONDARY OBJECTIVES:

I. To develop the infrastructure and strategy for a larger comparative intervention study (National Cancer Institute [NCI] R01).

OUTLINE: Participants are assigned to 1 of 2 arms.

ARM I: Participants receive standard post-treatment care consisting of regular cancer surveillance visits with treating oncologists.

ARM II: Participants complete survivorship care planning in close collaboration with treating oncologists.

After completion of study treatment, participants are followed up at 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage I, II, or III ovarian cancer
* Ability to read or understand English
* All subjects must have the ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

* Subjects, who in the opinion of the investigator, may not be able to comply with the safety monitoring requirements of the study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04-11; Primary Completion 2017-09-26 (Actual); Study Completion 2017-09-26 (Actual)

PRIMARY OUTCOMES:
Percentage of attrition | 2 months
  Descriptive statistics will be presented on those who agree to participate and the proportion of those approached who agree to participate. Descriptive statistics will also be presented for percentage of attrition (based on number of patients who failed to complete the 2 months study. Reasons for attrition will also be documented.
Total retention | 2 months
  Descriptive statistics will be presented for the total retention.
Recruitment rates | 2 months
  Important information regarding recruitment for the subsequent larger trial will be provided including estimates of the number of contacts needed to produce a qualified participant, the percentage of those who are qualified and agree to participate, and a retention rate.
Patient satisfaction assessed using the Survivor Satisfaction Tool and Debriefing Form | 2 months
  Quantitative and qualitative descriptive statistics will be analyzed using descriptive statistics and content analysis methods to determine satisfaction with the timing, content, and delivery of the intervention.

SECONDARY OUTCOMES:
Infrastructure for a larger comparative intervention study | 2 months
  The descriptive statistical estimates will be used for sample size determination for a larger subsequent study.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia Sun, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States